CLINICAL TRIAL: NCT04109248
Title: Clinical Pattern of Stroke and Transient Ischemic Attack Mimics in Patients Attending Neuropsychiatry Department in Assuit University Hospital
Brief Title: Clinical Pattern of Stroke and Transient Ischemic Attack Mimics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Loees Samir, Loees Samir Ishak, Assiut University
Other Study IDs: Stroke and TIA mimics
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
wide range of diagnoses may present like stroke, called stroke mimics as well as transient ischemic attacks .

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* aged above 18 years
* Accept all requirements of the study

Exclusion Criteria:

.Refuse participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient presented with an acute neurological symptom or focal neurological deficit that lasted for few minutes up to 24 hours or more in Neuropsychiatry department will be included in the study . These patients will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
True estimation of frequency of stroke and TIA mimics in patients attending Neuropsychiatry department in Assuit University Hospital. | 1 year
  frequency of stroke and TIA mimics in patients attending Neuropsychiatry department in Assuit University Hospital.